CLINICAL TRIAL: NCT04454853
Title: A Research of Value of Free Methylated DNA Detect in Lung Cancer on the Diagnosis and Treatment of Paraneoplastic Syndrome of Nervous System
Brief Title: Methylated DNA Detect in Paraneoplastic Syndrome of Nervous System
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUTH2017351
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Paraneoplastic Neurological Syndrome
Keywords: Paraneoplastic neurological syndrome; Cell-free DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lung cancer with positive methylated DNA: Blood DNA methylation abnormalities are found in lung cancer.
  Interventions: Other: Lung cancer; Other: Positive methylated DNA
- Lung cancer with negative methylated DNA: Blood DNA methylation abnormalities are not found in lung cancer.
  Interventions: Other: Lung cancer
- Suspected lung cancer with positive methylated DNA: Blood DNA methylation abnormalities are found in suspected lung cancer.
  Interventions: Other: Suspected lung cancer; Other: Positive methylated DNA
- Suspected lung cancer with negative methylated DNA: Blood DNA methylation abnormalities are not found in suspected lung cancer.
  Interventions: Other: Suspected lung cancer

INTERVENTIONS:
Other: Lung cancer — Paraneoplastic neurological syndrome (PNS) is a clinical syndrome that affects the central nervous system, peripheral nerves, neuromuscular junctions and muscles by the distant influence of the tumor. No tumor cells are visible at the neuropathy site.
  Groups: Lung cancer with negative methylated DNA; Lung cancer with positive methylated DNA
Other: Suspected lung cancer — Paraneoplastic neurological syndrome (PNS) is a clinical syndrome that affects the central nervous system, peripheral nerves, neuromuscular junctions and muscles by the distant influence of the tumor. No tumor cells are visible at the neuropathy site.
  Groups: Suspected lung cancer with negative methylated DNA; Suspected lung cancer with positive methylated DNA
Other: Positive methylated DNA — Tumor-free DNA (cfDNA) methylation detection is to determine the cancer condition and cancer type of the subject by detecting the methylation of free DNA released by tumor cells.
  Groups: Lung cancer with positive methylated DNA; Suspected lung cancer with positive methylated DNA

SUMMARY:
The purpose of this study is to verify whether the cell-free DNA of lung cancer in the blood can be used as a biomarker for early diagnosis and prognosis evaluation of patient with paraneoplastic syndrome of the nervous system.

DETAILED DESCRIPTION:
Paraneoplastic neurological syndrome (PNS) is a clinical syndrome that affects the central nervous system, peripheral nerves, neuromuscular junctions and muscles by the distant influence of the tumor. No tumor cells are visible in the neuropathy. The disease is a rare clinical syndrome, and lung cancer is the most common type of tumor that causes PNS.If PNS can be diagnosed when there are no tumor symptoms, not only can the cause of PNS be identified, but early tumors can be found for treatment time, and measures can be taken in the early stages of the tumor to improve survival. Tumor free DNA (cell-free DNA, cfDNA) methylation detection is to determine the cancer condition and cancer type of the subject by detecting the methylation of free DNA released by tumor cells. In normal cells, tumor suppressor genes are expressed and proto-oncogenes are silenced; in tumor cells, tumor suppressor genes are hypermethylated and silenced, and oncogenes are hypomethylated and activated. The release of free DNA into the blood will be quickly cleared in tens of minutes to several hours, which can reflect the body's cell damage in real time, and is of great significance for monitoring the early occurrence and development of the disease. At present, the sensitivity of lung cancer cf-DNA detection technology is close to 100%, and the specificity is 94%, which is an effective detection technology for early detection of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* The agnogenic typical neurological syndromes (including encephalomyelitis, marginal encephalitis, subacute cerebellar degeneration, strabismus ocular clonic-myoclonus, subacute sensory neuron disease, Lambert-Eaton myasthenic syndrome, skin Myositis, etc.) patient who predisposed to a tumor.
* Pathologically confirmed as lung cancer or suggested as lung cancer patient by imaging (pulmonary CT/Positron Emission Tomography-CT), tumor biomarkers, anti-brain tissue antibodies, etc.

Exclusion Criteria:

* Lacunar infarction
* Aortic atherosclerotic cerebral infarction
* Clear cardiogenic cerebral infarction
* Other related system diseases (arteritis, vascular dissection, migraine and vasospasm, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We recruited consecutive patients with paraneoplastic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Level of cf-DNA | 1 year after recruitment
  Tumor-free DNA (cfDNA) methylation detection is to determine the cancer condition and cancer type of the subject by detecting the methylation of free DNA released by tumor cells.

SECONDARY OUTCOMES:
Changes of mRS score | 1 year after recruitment
  Documentation in the medical record of a Modified Rankin Score (mRS). The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. Standardized interviews to obtain a mRS score are recommended at 3 months (90 days) following hospital discharge.
Survival time | 1 years after recruitment
  The time interval from disease diagnosis to death
1-year mortality rate | 1 year after recruitment
  The rate of death among all the inclusion patients after 1 year
Incidence of lung cancer | 1 year after recruitment
  The rate of lung cancer occurence among all the inclusion patients

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No